CLINICAL TRIAL: NCT06340373
Title: Clinical & Angiographic Outcomes of Drug-coated Balloon Angioplasty After Successful Revascularization of Native Coronary Lesions
Brief Title: Clinical and Angiographic Outcomes of Post-drug-coated Balloon Angioplasty in Native Coronary Lesions
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Bangladesh (Other)
Responsible Party: Principal Investigator, Mohsin Ahmed, Professor, National Institute of Cardiovascular Diseases, Bangladesh
Other Study IDs: NICVD/ 2023/ 32; NICVD /Ethical/ 2023/ 32 (Other: National Institute of Cardiovascular Diseases(NICVD))
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty; Balloon Angioplasty; Native Coronary Lesions; Coronary Artery Disease; Bangladesh
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with native coronary lesions (2.0-3.5 mm diameter) after drug-coated balloon angioplasty: Patients with successful revascularization of native coronary lesions (diameter >2.0 mm and ≦3.5 mm at visual estimation) by drug-coated balloon angioplasty and follow up after six month by coronary angiography
  Interventions: Device: DCB Angioplasty

INTERVENTIONS:
Device: DCB Angioplasty — Drug-coated balloons (DCB) are designed to deliver drugs (antiproliferative drugs: Paclitaxel, Sirolimus etc.) to the target lesion/vessel wall without leaving nothing behind unlike stent strut or drug delivery system. Drug coated balloons (DCB) allow the homogenous transfer of an anti-proliferative drug to reduce neo-intimal hyperplasia whilst maintaining normal vessel anatomy and function

SUMMARY:
The progression of cardiac revascularization techniques, starting with standard balloon angioplasty (POBA) and progressing to the creation of drug-coated balloons (DCB) and drug-eluting stents (DES). The study's justification is presented, with a focus on the significance of comprehending the clinical and angiographic outcomes of DCB angioplasty, especially when considering the Bangladeshi population.

This study's main goal is to observe the clinical and angiographic outcomes of drug-coated balloon angioplasty after native coronary lesions that have been successfully revascularized. A few specific goals are to evaluate angiographic results (like percentage diameter stenosis, vascular remodelling, restenosis, and thrombosis) after DCB angioplasty and to assess clinical outcomes (like worsening angina, target vessel MI, ischemia-driven TLR, and cardiac mortality).

This observational study will take place from January to December 2024 at the Department of Cardiology, National Institute of Cardiovascular Diseases. The study population will be individuals who had successful revascularization of native coronary lesions with DCB angioplasty six months before. The study includes non-randomized purposive sampling, and the sample size will be determined by drawing on previous studies.

Every patient will receive a thorough clinical assessment that includes a history, physical examination, electrocardiogram, and biochemical testing. The data will be analysed in accordance with the assessment of angiographic outcomes by follow-up angiography.

The purpose of this study is to give useful insights into the clinical and angiographic results of DCB angioplasty in Bangladeshi patients with native coronary lesions, including the growing body of knowledge on the efficacy and safety of this therapeutic strategy in specific populations.

DETAILED DESCRIPTION:
In recent years, drug-coated balloon (DCB) therapy has been rapidly accepted in clinical practice, especially for the treatment of in-stent restenosis. More recently, the use of DCB is spreading to de novo CAD. The DCB has beneficial features, such as allowing local drug delivery without the need to implant any metal. Subsequently, the duration of dual antiplatelet therapy (DAPT) is shortened. Importantly, the DCB is just a delivery vehicle, and does not assist in dilating narrowed coronary vessels. Thus, lesion preparation with standard balloon angioplasty is the key to successful DCB treatment, and is essential before the use of a DCB. The aim of effective lesion preparation is to gain sufficient luminal enlargement, while minimizing coronary dissection. As DCBs are fulfilling the concept of "leaving nothing behind" and guidelines are also recommended as class I indication the use of DCBs have become an alternative therapeutic option for the treatment of ISR & small de novo vessel. Till to date no such type of study conducted in Bangladesh. That's why the investigators designed this study with the aim to observe clinical and angiographic outcomes of drug-coated balloon angioplasty after successful revascularization of native coronary lesions among Bangladeshi population which is very essential and relevant in the context of Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients with successful revascularization of native coronary lesions (diameter >2.0 mm and ≦3.5 mm at visual estimation) six months back by drug-coated balloon angioplasty.
* Informed consent to participate in the study

Exclusion Criteria:

* Creatinine clearance <30 ml/min
* Left ventricular ejection fraction <30%
* Life expectancy <12 months
* Target lesion/vessel with any of the following characteristics: - concomitant PCI at the same vessel with any device (vessels are considered: left anterior descending, circumflex or right coronary artery)
* Previous stent implantation at target vessel (left anterior descending artery; circumflex artery; right coronary artery)
* Patient who will not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with successful revascularization of native coronary lesions (diameter >2.0 mm and ≦3.5 mm at visual estimation) six months back by drug-coated balloon angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
CCS (Canadian Cardiovascular Society) Class of Worsening angina of each participant | Six months
  Exacerbation of chest pain symptoms following the procedure, possibly indicating complications or inadequate treatment effectiveness.
Number of participants with target vessel Myocardial infarction | Six months
  Potential damage to the heart muscle due to reduced blood flow in the treated vessel, possibly resulting from a clot or other factors related to the procedure.
Ischemia-driven Target lesion revascularization (TLR) each participant | Six months
  The need for repeat intervention (such as another angioplasty or stent placement) in the same artery that was initially treated with the drug-coated balloon.
Occurrence of Cardiac death in the participants | Six months
  The occurrence of death directly related to a cardiac event following the procedure. This outcome indicates a severe complication possibly stemming from factors such as acute myocardial infarction, arrhythmias, or other cardiovascular complications directly impacting the heart's function and leading to fatal consequences.
Site of the lesion | Six months
  Vessel & Location
Lesion Length | Six months
  < 10 mm/ 10-20/ > 20 mm
% of Stenosis | Six months
  Before / After 6 months
Thrombolysis in Myocardial Infarction (TIMI) Flow | Six months
  Before / After 6 months
Pre dilatation - Balloon Type | Six months
  1. Non-compliant/ Semi compliant/ Compliant.
  2. Balloon size -
  3. Pressure -

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Mohsin Ahmed, MD, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of CardioVascular Diseases, Dhaka, Bangladesh

REFERENCES:
- [Background] Brami P, Fischer Q, Pham V, Seret G, Varenne O, Picard F. Evolution of Coronary Stent Platforms: A Brief Overview of Currently Used Drug-Eluting Stents. J Clin Med. 2023 Oct 24;12(21):6711. doi: 10.3390/jcm12216711. PMID 37959177
- [Background] Bravo Baptista S. The third generation of drug-eluting stents: Reassuring data while we wait for the next one. Rev Port Cardiol (Engl Ed). 2021 Feb;40(2):77-80. doi: 10.1016/j.repc.2020.12.004. Epub 2020 Dec 25. No abstract available. English, Portuguese. PMID 33358574
- [Background] Jackson D, Tong D, Layland J. A review of the coronary applications of the drug coated balloon. Int J Cardiol. 2017 Jan 1;226:77-86. doi: 10.1016/j.ijcard.2016.09.045. Epub 2016 Sep 16. PMID 27792992
- [Background] Indermuehle A, Bahl R, Lansky AJ, Froehlich GM, Knapp G, Timmis A, Meier P. Drug-eluting balloon angioplasty for in-stent restenosis: a systematic review and meta-analysis of randomised controlled trials. Heart. 2013 Mar;99(5):327-33. doi: 10.1136/heartjnl-2012-302945. Epub 2013 Jan 18. PMID 23335497
- [Background] Scheller B, Clever YP, Kelsch B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Speck U, Bohm M, Cremers B. Long-term follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. JACC Cardiovasc Interv. 2012 Mar;5(3):323-30. doi: 10.1016/j.jcin.2012.01.008. PMID 22440499
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Ong PJ, Zeymer U, Waliszewski M, Tan J, Ho HH. Differences in clinical and angiographic profiles between Asian and Western patients with coronary artery disease: insights from the prospective "real world" paclitaxel-coated balloon registry. Int J Cardiol. 2014 Jul 15;175(1):199-200. doi: 10.1016/j.ijcard.2014.04.239. Epub 2014 Apr 28. No abstract available. PMID 24820752
- [Background] Akiyama T, Moussa I, Reimers B, Ferraro M, Kobayashi Y, Blengino S, Di Francesco L, Finci L, Di Mario C, Colombo A. Angiographic and clinical outcome following coronary stenting of small vessels: a comparison with coronary stenting of large vessels. J Am Coll Cardiol. 1998 Nov 15;32(6):1610-8. doi: 10.1016/s0735-1097(98)00444-6. PMID 9822086
- [Background] Her AY, Shin ES, Bang LH, Nuruddin AA, Tang Q, Hsieh IC, Hsu JC, Kiam OT, Qiu C, Qian J, Ahmad WAW, Ali RM. Drug-coated balloon treatment in coronary artery disease: Recommendations from an Asia-Pacific Consensus Group. Cardiol J. 2021;28(1):136-149. doi: 10.5603/CJ.a2019.0093. Epub 2019 Sep 30. PMID 31565793
- [Background] Pan L, Lu W, Han Z, Pan S, Wang X, Shan Y, Wang X, Zheng X, Li R, Zhou Y, Qin P, Shi Q, Zhou S, Zhang W, Guo S, Zhang P, Qin X, Sun G, Qin Z, Huang Z, Qiu C. Clinical outcomes of drug-coated balloon in coronary lesions: a real-world, all-comers study. Clin Res Cardiol. 2022 Jul;111(7):732-741. doi: 10.1007/s00392-021-01895-y. Epub 2021 Jul 27. PMID 34313800